CLINICAL TRIAL: NCT01140451
Title: A Phase 3 Extension Study of Ataluren (PTC124®) in Subjects With Nonsense-Mutation-Mediated Cystic Fibrosis
Brief Title: Extension Study of Ataluren (PTC124) in Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-009e-CF; Orphan Product Grant #FD003715 (Other Grant/Funding Number: FDA Office of Orphan Products Development (OOPD)); 2010-019692-30 (EudraCT Number)
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ataluren

STUDY DESIGN:
Masking Description: This extension study was not blinded. The investigators and participants remained blinded to the Study 009 treatment assignments throughout participation in Study PTC124-GD-009e-CF.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ataluren/Ataluren (Experimental): Participants who received double-blind ataluren during Study 009 will continue to receive open-label ataluren 3 times per day TID: 10 milligram (mg)/kilogram (kg) of body weight with breakfast, 10 mg/kg with lunch, and 20 mg/kg with dinner (total dose 40 mg/kg/day), for up to 96 weeks. Participants will be followed for 4 weeks after treatment.
  Interventions: Drug: Ataluren
- Placebo/Ataluren (Experimental): Participants who received double-blind placebo during Study 009 will receive open-label ataluren TID: 10 mg/kg of body weight with breakfast, 10 mg/kg with lunch, and 20 mg/kg with dinner (total dose 40 mg/kg/day), for up to 96 weeks. Participants will be followed for 4 weeks after treatment.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Ataluren will be provided as a vanilla-flavored powder to be mixed with water or milk.
  Other Names: PTC124

SUMMARY:
Cystic fibrosis (CF) is a genetic disorder caused by a mutation in the gene that makes the cystic fibrosis transmembrane conductance regulator (CFTR) protein. A specific type of mutation called a nonsense (premature stop codon) mutation is the cause of CF in approximately 10% of patients with the disease. Ataluren is an orally delivered investigational drug that has the potential to overcome the effects of the nonsense mutation. This study is a Phase 3 extension trial that will evaluate the long-term safety of ataluren in adult and pediatric participants with nonsense mutation CF (nmCF), as determined by adverse events and laboratory abnormalities. The study will also assess changes in pulmonary function, CF pulmonary exacerbations, health-related quality of life, antibiotic use for CF-related infections, CF-related disruptions to daily living, body weight, and CF pathophysiology. Funding source for this study is the FDA OOPD.

DETAILED DESCRIPTION:
This Phase 3, open-label, safety and efficacy study will be performed at sites in North America, Europe, and Israel. The study will enroll up to approximately 208 participants with nmCF who participated in a previous Phase 3 study of ataluren (PTC124-GD-009-CF [Study 009], NCT00803205). Participants will receive study drug 3 times per day (TID) (at breakfast, lunch, and dinner) for approximately 48 weeks (approximately 1 year). Study assessments will be performed at clinic visits every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Completion of blinded study drug treatment in the previous Phase 3 study (PTC124-GD-009-CF).
* Ability to provide written informed consent (parental/guardian consent if applicable)/assent (if <18 years of age).
* In participants who are sexually active, willingness to abstain from sexual intercourse or employ a barrier or medical method of contraception during ataluren administration and the 4-week follow up period.
* Willingness and ability to comply with scheduled visits, drug administration plan, study procedures, laboratory tests, and study restrictions.

Exclusion Criteria:

* Known hypersensitivity to any of the ingredients or excipients of the study drug (list provided at study sites).
* Current pregnancy or lactating, or pregnancy or lactating during the previous Phase 3 study.
* Ongoing participation in any other therapeutic clinical trial.
* Prior or ongoing medical condition (for example, concomitant illness, psychiatric condition, behavioral disorder, alcoholism, drug abuse), medical history, physical findings, ECG findings, or laboratory abnormality that, in the Investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of treatment or follow up would be completed, or could impair the assessment of study results.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2010-08-12 (Actual); Primary Completion 2013-12-02 (Actual); Study Completion 2013-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Temitayo Ajayi, MD, Study Director — PTC Therapeutics, Inc.
Locations (31):
- United States (15):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Miller Children's Hospital Long Beach, Long Beach, California
  - Lucile Packard Children's Hospital, Palo Alto, California
  - The Children's Hospital, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Emory University Cystic Fibrosis Center, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - St. Vincent's Hospital, New York, New York
  - New York Medical College, Valhalla, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
- Belgium (4):
  - Hôpital Erasme, Brussels
  - Hôpital Universitaire des Enfants Reine Fabiola, Brussels
  - University Hospital Brussels, Brussels
  - University Hospital Leuven, Leuven
- University of Toronto, Toronto, Canada
- France (3):
  - Hôpital Cochin, Paris
  - Hôpital Necker - Enfants Malades, Paris
  - Hôpital des Enfants, Toulouse
- Klinikum der Universität Köln, Cologne, Germany
- Hadassah University Hospital - Mount Scopus, Jerusalem, Israel
- Italy (2):
  - Università La Sapienza, Roma
  - Azienda Ospedaliera di Verona, Verona
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Hospital Universitario La Paz, Madrid, Spain
- Karolinska University Hospital, Huddinge, Stockholm, Sweden
- Belfast City Hospital, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PTC Therapeutics, Inc. website — http://www.ptcbio.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, open-label extension study of the safety and efficacy of ataluren in male and female participants with nonsense mutation cystic fibrosis (nmCF) aged ≥6 years who successfully completed Study PTC124-GD-009-CF (NCT00803205 [Study 009]).
Pre-assignment Details: Participants began the open-label extension study immediately after completing end-of-study visit (Week 48) in Study 009 to avoid interruption in treatment. Most assessments performed at Study 009's final visit were used as Baseline assessments in Study PTC124-GD-009e-CF (009e). Investigators and participants remained blinded to Study 009 dosing.
Groups:
- Ataluren/Ataluren: Participants who received double-blind ataluren during Study 009 continued to receive open-label ataluren taken 3 times per day (TID): 10 milligram (mg)/kilogram (kg) of body weight with breakfast, 10 mg/kg with lunch, and 20 mg/kg with dinner (total dose 40 mg/kg/day), for up to 96 weeks. Participants were followed for 4 weeks after treatment.
- Placebo/Ataluren: Participants who received double-blind placebo during Study 009 received open-label ataluren TID: 10 mg/kg of body weight with breakfast, 10 mg/kg with lunch, and 20 mg/kg with dinner (total dose 40 mg/kg/day), for up to 96 weeks. Participants were followed for 4 weeks after treatment.
Period: Overall Study
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Started (The first week of Study 009e was Total Study Week 48 for Studies 009 and 009e combined.) | 95 | 96
Completed 24 Weeks (Week 24 of Study 009e was Total Study Week 72) | 89 | 86
Completed 48 Weeks (Week 48 of Study 009e was Total Study Week 96) | 78 | 70
Completed 72 Weeks (Week 72 of Study 009e was Total Study Week 120) | 63 | 62
Completed 96 Weeks (Week 96 of Study 009e was Total Study Week 144) | 57 | 54
As-Treated Population (Received at least 1 dose of study drug in Study 009e) | 95 | 96
96-Week Completer Population (Completed 48 weeks of treatment in both Study 009 and Study 009e) | 78 | 70
144-Week Completer Population (Completed 48 weeks of treatment in Study 009 and 96 weeks in Study 009e) | 57 | 54
Completed (Study completion for Study 009e was Week 100 (Total Study Week 148)) | 57 | 54
Not Completed | 38 | 42
Not completed — Withdrawal by Subject | 26 | 33
Not completed — Adverse Event | 2 | 6
Not completed — Physician Decision | 5 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Participants Planning Pregnancy | 3 | 0

BASELINE CHARACTERISTICS:
Population: The Study 009e As-Treated Population: participants who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren | Total
Number analyzed (Participants) | 95 | 96 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.9 (10.04) | 24.9 (9.29) | 23.9 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 97
  Male | 47 | 47 | 94

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship that occurred or worsened in the period extending from the first dose of study drug to 6 weeks after the last dose of study drug. A serious adverse event (SAE) was an adverse event (AE) resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. AE severity was graded as follows: Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening; Grade 5: fatal. A TEAE was considered related if in the opinion of the Investigator it was possibly or probably caused by the study drug. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the Adverse Events module.
Time Frame: Baseline (Week 1 [Total Study Week 48]) up to 4 Weeks Post-Treatment (Week 100 [Total Study Week 148]) or Premature Discontinuation (PD) (whichever occurred first)
Population: The Study 009e As-Treated Population: participants who received at least 1 dose of study drug.
Measure: Number; unit: percent of participants
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
percent of participants
  At least 1 TEAE | 100 | 97.9
  Grade 1 TEAE | 14.7 | 18.8
  Grade 2 TEAE | 62.1 | 51.0
  Grade 3 TEAE | 23.2 | 26.0
  Grade 4 TEAE | 0 | 1.0
  Grade 5 TEAE | 0 | 1.0
  Unrelated TEAE | 29.5 | 26.0
  Unlikely related TEAE | 37.9 | 33.3
  Possibly related TEAE | 28.4 | 31.3
  Probably related TEAE | 4.2 | 7.3
  Discontinued due to TEAE | 2.1 | 6.3
  Serious TEAE | 50.5 | 57.3

2. Primary Outcome: Number of Participants With Any Treatment-Emergent Laboratory Abnormality (TELA)
Description: A TELA is any abnormal laboratory value that started or worsened after administration of study drug. Abnormal values were defined as values outside normal range. Values considered abnormal included -Hepatic: Serum total bilirubin ≥1.5*upper limit of normal (ULN); serum gamma glutamyl transferase >2.5*ULN; serum alanine aminotransferase increase of >150 units/liter (U/L) without increased creatine kinase; -Adrenal: plasma adrenocorticotropic hormone >ULN (normal cortisol); -Renal: serum cystatin C >1.33 milligrams (mg)/L; serum creatinine >ULN-1.5*ULN for age; serum blood urea nitrogen ≥1.5*ULN; urine protein:creatinine >0.40 mg/deciliter (dL):mg/dL; urine protein:osmolality >0.30 mg/L:milliosmoles/kilogram; urine blood 2+; - Serum Electrolytes: serum sodium >150 millimoles (mmol)/L, <130 mmol/L; serum potassium >5.5, <3.0 mmol/L; serum magnesium >1.23 mmol/L, <0.5 mmol/L; total serum calcium >2.9 mmol/L, <2.0 mmol/L; serum phosphorous <0.8 mmol/L; serum biocarbonate- <16 mmol/L.
Time Frame: Baseline (Week 1 [Total Study Week 48]) up to 4 Weeks Post-Treatment (Week 100 [Total Study Week 148]) or PD (whichever occurred first)
Population: The Study 009e As-Treated Population: participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
Participants
  Renal laboratory abnormality | 13 | 18
  Serum electrolyte laboratory abnormality | 39 | 47
  Hepatic laboratory abnormality | 44 | 49
  Adrenal laboratory abnormality | 5 | 3

3. Secondary Outcome: Percentage of Predicted Function (Percent-Predicted) of Forced Expiratory Volume in 1 Second (FEV1) at Baseline
Description: Spirometry was used to assess pulmonary function by measuring the percent-predicted, which was determined on the basis of the height value obtained at the same study visit, for FEV1 (the amount of air that can be exhaled in 1 second). Spirometry was validated by using current guidelines of the American Thoracic Society (ATS) and European Respiratory Society (ERS). Baseline was defined as Week 1 or the most recent value of percent-predicted FEV1 prior to the first dose of open-label treatment in Study 009e.
Time Frame: Baseline (Week 1 [Total Study Week 48])
Population: The Study 009e As-Treated Population: participants who received at least 1 dose of study drug. Here, 'Number Analyzed' signifies participants evaluable for the specified week.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
percentage of predicted FEV1 | 60.61 (17.075) | 56.49 (15.954)

4. Secondary Outcome: Percentage Change From Baseline in Percent-Predicted of FEV1 at Weeks 48 and 96
Description: Spirometry was used to assess pulmonary function by measuring the percent-predicted, which was determined on the basis of the height value obtained at the same study visit, for FEV1 (the amount of air that can be exhaled in 1 second). Spirometry was validated by using current guidelines of the American Thoracic Society (ATS) and European Respiratory Society (ERS). The percentage of change in percent-predicted of FEV1 was calculated as follows: ((percent-predicted FEV1-Baseline percent-predicted FEV1)/Baseline percent-predicted FEV1)*100. Baseline was defined as Week 1 or the most recent value of percent-predicted FEV1 prior to the first dose of open-label treatment in Study 009e. A positive change from Baseline indicates that FEV1 improved.
Time Frame: Week 48 (Total Study Week 96), End of Treatment (EOT) (Week 96 [Total Study Week 144])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
percent change
  Change From Baseline at Week 48: number analyzed (Participants) | 75 | 66
  Change From Baseline at Week 48 | -0.73 (12.170) | 1.09 (23.025)
  Change From Baseline at Week 96: number analyzed (Participants) | 55 | 50
  Change From Baseline at Week 96 | -3.09 (12.304) | -2.12 (16.893)

5. Post Hoc Outcome: Percent-Predicted of FEV1 in the 96-Week Completer Population at Baseline
Description: Spirometry was used to assess pulmonary function by measuring the percent-predicted, which was determined on the basis of the height value obtained at the same study visit, for FEV1 (the amount of air that can be exhaled in 1 second). Spirometry was validated by using current guidelines of the ATS and ERS. Analyses with the Completer populations were performed to complement the analyses of the Study 009e As-Treated population. Baseline was defined as Week 1 or the most recent value of percent-predicted FEV1 prior to the first dose of open-label treatment in Study 009e.
Time Frame: Baseline (Week 1 [Total Study Week 48])
Population: Study 009/009e 96-Week Completer Population: participants who completed 48 weeks of treatment with ataluren or placebo in Study 009 and at least 48 weeks of treatment with ataluren in Study 009e. Here, 'Number Analyzed' signifies participants evaluable for the specified week.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 78 | 70
percentage of predicted FEV1 | 60.89 (13.320) | 59.50 (15.622)

6. Post Hoc Outcome: Percentage Change From Baseline in Percent-Predicted of FEV1 in the 96-Week Completer Population Over a Total of 96 Weeks of Treatment
Description: Spirometry was used to assess pulmonary function by measuring the percent-predicted, which was determined on the basis of the height value obtained at the same study visit, for FEV1 (the amount of air that can be exhaled in 1 second). Spirometry was validated by using current guidelines of the ATS and ERS. The percentage of change in percent-predicted of FEV1 was calculated as follows: ((percent-predicted FEV1-Baseline percent-predicted FEV1)/Baseline percent-predicted FEV1)*100. Analyses with the Completer populations were performed to complement the analyses of the Study 009e As-Treated population. Baseline was defined as Week 1 or the most recent value of percent-predicted FEV1 prior to the first dose of open-label treatment in Study 009e. A positive change from Baseline indicates that FEV1 improved.
Time Frame: Week 48 (Total Study Week 96)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 78 | 70
percent change | -1.63 (13.239) | -5.13 (12.061)

7. Post Hoc Outcome: Percent-Predicted of FEV1 in the 144-Week Completer Population at Baseline
Description: as for outcome 5
Time Frame: Baseline (Week 1 [Total Study Week 48])
Population: Study 009/009e 144-Week Completer Population: participants who completed 48 weeks of treatment with ataluren or placebo in Study 009 and at least 96 weeks of treatment with ataluren in Study 009e. Here, 'Number Analyzed' signifies participants evaluable for the specified week.
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 57 | 54
percentage of predicted FEV1 | 61.68 (13.790) | 60.28 (16.202)

8. Post Hoc Outcome: Percentage Change From Baseline in Percent-Predicted of FEV1 in the 144-Week Completer Population Over a Total of 144 Weeks of Treatment
Description: as for outcome 6
Time Frame: EOT (Week 96 [Total Study Week 144])
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 57 | 54
percent change | -3.69 (16.068) | -5.89 (14.854)

9. Secondary Outcome: Percent-Predicted of Forced Vital Capacity (FVC) at Baseline
Description: Spirometry was used to assess pulmonary function by measuring the percent-predicted, which was determined on the basis of the height value obtained at the same study visit, for FVC (the amount of air that can be exhaled after taking a deep breath). Spirometry was validated by using current guidelines of the ATS and ERS. Baseline was defined as Week 1 or the most recent value of percent-predicted FVC prior to the first dose of open-label treatment in Study 009e.
Time Frame: Baseline (Week 1 [Total Study Week 48])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of predicted FVC
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
percentage of predicted FVC | 76.37 (15.254) | 73.26 (14.133)

10. Secondary Outcome: Percentage Change From Baseline in Percent-Predicted of FVC at Weeks 48 and 96
Description: Spirometry was used to assess pulmonary function by measuring the percent-predicted, which was determined on the basis of the height value obtained at the same study visit, for FVC (the amount of air that can be exhaled after taking a deep breath). Spirometry was validated by using current guidelines of the ATS and ERS. The percentage of change in percent-predicted of FVC was calculated as follows: ((percent-predicted FVC-Baseline percent-predicted FVC)/Baseline percent-predicted FVC)*100. Baseline was defined as Week 1 or the most recent value of percent-predicted FVC prior to the first dose of open-label treatment in Study 009e. A positive change from Baseline indicates that FVC improved.
Time Frame: Week 48 (Total Study Week 96), EOT (Week 96 [Total Study Week 144])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
percent change
  Change From Baseline at Week 48: number analyzed (Participants) | 75 | 66
  Change From Baseline at Week 48 | 0.05 (10.690) | 0.69 (15.658)
  Change From Baseline at Week 96: number analyzed (Participants) | 55 | 50
  Change From Baseline at Week 96 | -1.48 (11.080) | -1.17 (13.940)

11. Secondary Outcome: Percent-Predicted of Forced Expiratory Flow Between 25% and 75% of Expiration (FEF25-75) at Baseline
Description: Spirometry was used to assess pulmonary function by measuring the percent-predicted, which was determined on the basis of the height value obtained at the same study visit, for FEF25-75 (the rate of air flow during the middle part of an exhalation). Spirometry was validated by using current guidelines of the ATS and ERS. Baseline was defined as Week 1 or the most recent value of percent-predicted FEF25-75 prior to the first dose of open-label treatment in Study 009e.
Time Frame: Baseline (Week 1 [Total Study Week 48])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of predicted FEF25-75
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
percentage of predicted FEF25-75 | 38.16 (24.594) | 33.11 (23.775)

12. Secondary Outcome: Percentage Change From Baseline in Percent-Predicted of FEF25-75 at Weeks 48 and 96
Description: Spirometry was used to assess pulmonary function by measuring the percent-predicted, which was determined on the basis of the height value obtained at the same study visit, for FEF25-75 (the rate of air flow during the middle part of an exhalation). Spirometry was validated by using current guidelines of the ATS and ERS. The percentage of change in percent-predicted of FEF25-75 was calculated as follows: ((percent-predicted FEF25-75-Baseline percent-predicted FEF25-75)/Baseline percent-predicted FEF25-75)*100. Baseline was defined as Week 1 or the most recent value of percent-predicted FEF25-75 prior to the first dose of open-label treatment in Study 009e. A positive change from Baseline indicates that FEF25-75 improved.
Time Frame: Week 48 (Total Study Week 96), EOT (Week 96 [Total Study Week 144])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
percent change
  Change From Baseline at Week 48: number analyzed (Participants) | 75 | 66
  Change From Baseline at Week 48 | -0.55 (22.447) | 7.89 (58.780)
  Change From Baseline at Week 96: number analyzed (Participants) | 55 | 50
  Change From Baseline at Week 96 | -5.55 (24.043) | -3.29 (25.283)

13. Secondary Outcome: Number of Participants With Pulmonary Exacerbations as Defined by Modified Fuch's Criteria
Description: A Respiratory Event Form (REF), which collected data on various signs, symptoms, and effects for each event, was completed by the Investigator when informed by the participant of a respiratory event. Pulmonary exacerbations were assessed by using the modified Fuchs' criteria, which defines an exacerbation as a respiratory event requiring treatment with parenteral antibiotics for any 4 of the following 12 symptoms with or without intravenous (IV) antibiotics: change in sputum; new or increased hemoptysis; increased cough; increased dyspnea; fatigue; temperature >38°C; anorexia; sinus pain; change in sinus discharge; change in physical examination of the chest; or decrease in pulmonary function by 10% or more from a previously recorded value; or radiographic changes indicative of pulmonary function.
Time Frame: Baseline (Week 1 [Total Study Week 48]) up to Week 48 and EOT (Week 96) (Total Study Weeks 96 and 144)
Population: The Study 009e As-Treated Population: participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
Participants
  Week 1 up to Week 48 | 50 | 56
  Week 1 up to Week 96 | 57 | 68

14. Secondary Outcome: Rate of Pulmonary Exacerbations as Defined by Modified Fuch's Criteria Over 48 Weeks
Description: A REF, which collected data on various signs, symptoms, and effects for each event, was completed by the Investigator when informed by the participant of a respiratory event. Pulmonary function was assessed by using the modified Fuchs' criteria, which defines an exacerbation as a respiratory event requiring treatment with parenteral antibiotics for any 4 of the following 12 symptoms with or without treatment with IV antibiotics: change in sputum; new or increased hemoptysis; increased cough; increased dyspnea; fatigue; temperature >38°C; anorexia; sinus pain; change in sinus discharge; change in physical examination of the chest; decrease in pulmonary function by 10% or more from a previously recorded value; or radiographic changes indicative of pulmonary function. The 48-week exacerbation rate was determined by adding the weekly rates for each arm for each 48-week period and dividing the sum by 48.
Time Frame: Baseline (Week 1 [Total Study Week 48]) up to Week 48 (Total Study Week 96)
Population: The Study 009e As-Treated Population: participants who received at least 1 dose of study drug.
Measure: Mean (95% Confidence Interval); unit: exacerbations
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
exacerbations | 1.150 [0.843 to 1.457] | 1.614 [1.163 to 2.064]

15. Secondary Outcome: Duration of Pulmonary Exacerbations as Defined by Modified Fuch's Criteria
Description: A REF, which collected data on various signs, symptoms, and effects for each event, was completed by the Investigator when informed by the participant of a respiratory event. Pulmonary function was assessed by using the modified Fuchs' criteria, which defines an exacerbation as a respiratory event requiring treatment with parenteral antibiotics for any 4 of the following 12 symptoms with or without treatment with IV antibiotics: change in sputum; new or increased hemoptysis; increased cough; increased dyspnea; fatigue; temperature >38°C; anorexia; sinus pain; change in sinus discharge; change in physical examination of the chest; decrease in pulmonary function by 10% or more from a previously recorded value; or radiographic changes indicative of pulmonary function. Duration over a 5-week interval is presented. The duration was calculated as follows: estimated date of return to a stable state (as determined by the Investigator) - estimated date of onset of symptoms.
Time Frame: Weeks 43 up to 48 and Weeks 91 up to 96 (Total Study Weeks 91 up to 96 and Weeks 139 up to 144)
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
days
  Week 43 up to Week 48: number analyzed (Participants) | 80 | 79
  Week 43 up to Week 48 | 3.675 [1.394 to 5.956] | 4.734 [2.258 to 7.210]
  Week 91 up to Week 96: number analyzed (Participants) | 60 | 57
  Week 91 up to Week 96 | 3.567 [1.124 to 6.010] | 3.912 [1.742 to 6.083]

16. Secondary Outcome: Number of Participants With Severe Pulmonary Exacerbations as Defined by Modified Fuch's Criteria
Description: A REF, which collected data on various signs, symptoms, and effects for each event, was completed by the Investigator when informed by the participant of a respiratory event. Pulmonary function was assessed by using the modified Fuchs' criteria, which defines an exacerbation as a respiratory event requiring treatment with parenteral antibiotics for any 4 of the following 12 symptoms with or without treatment with IV antibiotics: change in sputum; new or increased hemoptysis; increased cough; increased dyspnea; fatigue; temperature >38°C; anorexia; sinus pain; change in sinus discharge; change in physical examination of the chest; decrease in pulmonary function by 10% or more from a previously recorded value; or radiographic changes indicative of pulmonary function. Severity of pulmonary exacerbations over a 5-week interval is presented. The severity of pulmonary exacerbations were graded as mild, moderate, or severe.
Time Frame: Weeks 43 up to 48 and Weeks 91 up to 96 (Total Study Weeks 91 up to 96 and Weeks 139 up to 144)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
Participants
  Week 43 up to Week 48: number analyzed (Participants) | 71 | 73
  Week 43 up to Week 48 | 1 | 1
  Week 91 up to Week 96: number analyzed (Participants) | 53 | 49
  Week 91 up to Week 96 | 0 | 1

17. Secondary Outcome: Change From Baseline for the Respiratory Domain Score of the Cystic Fibrosis (CF) Questionnaire-Revised (CFQ-R) at Weeks 48 and 96
Description: The CFQ-R consists of 44 items, including generic scales of physical functioning, role functioning, vitality, health perceptions, emotional functioning, and social functioning, and CF-specific scales of respiratory and digestive symptoms, body image, eating disturbances, and treatment burden. Questions are scored on a scale from 1 to 4, with higher scores indicating better quality of life (QOL). For some questions, the scale was reversed, so that 1 indicated better QOL. Domain scores were linearly transformed to a 0-100 scale, so that higher scores indicate better QOL. Domain scores were calculated by using the following formula: 100 * (sum of responses - minimum possible sum)/ (maximum possible sum - minimum possible sum). The minimum possible sum = number of questions * 1; the maximum possible = the number of questions * 4. Baseline was Week 1. A negative change from Baseline indicates that health has worsened. Participants may have switched age groups during the study.
Time Frame: Baseline (Week 1 [Total Study Week 48]), Week 48 (Total Study Week 96), EOT (Week 96 [Total Study Week 144])
Population: The Study 009e As-Treated Population: participants who received at least 1 dose of study drug. Here, 'Number Analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
units on a scale
  Aged 6-11 years, Baseline: number analyzed (Participants) | 8 | 3
  Aged 6-11 years, Baseline | 83.333 (8.9087) | 86.111 (17.3472)
  Aged 6-11 years, Change From Baseline at Week 48: number analyzed (Participants) | 7 | 3
  Aged 6-11 years, Change From Baseline at Week 48 | -13.095 (19.7538) | -0 (0)
  Aged 6-11 years, Change From Baseline at Week 96: number analyzed (Participants) | 6 | 1
  Aged 6-11 years, Change From Baseline at Week 96 | -5.556 (10.0922) | 0 (NA) — Standard deviation cannot be calculated with an N of 1.
  Aged 12-13 years, Baseline: number analyzed (Participants) | 6 | 3
  Aged 12-13 years, Baseline | 75.000 (16.6667) | 63.889 (4.8113)
  Aged 12-13 years, Change From Baseline at Week 48: number analyzed (Participants) | 2 | 2
  Aged 12-13 years, Change From Baseline at Week 48 | 0 (11.7851) | 16.667 (0)
  Aged 12-13 years, Change From Baseline at Week 96: number analyzed (Participants) | 0 | 0
  Age ≥14 years, Baseline: number analyzed (Participants) | 80 | 90
  Age ≥14 years, Baseline | 66.181 (20.5449) | 65.123 (18.1322)
  Age ≥14 years, Change From Baseline at Week 48: number analyzed (Participants) | 64 | 64
  Age ≥14 years, Change From Baseline at Week 48 | 2.691 (17.4280) | 3.819 (16.2311)
  Age ≥14 years, Change From Baseline at Week 96: number analyzed (Participants) | 43 | 51
  Age ≥14 years, Change From Baseline at Week 96 | 5.039 (16.4811) | 1.307 (20.9228)
  All participants, Baseline: number analyzed (Participants) | 94 | 96
  All participants, Baseline | 68.203 (20.1408) | 65.567 (18.1927)
  All participants, Change From Baseline at Week 48: number analyzed (Participants) | 77 | 70
  All participants, Change From Baseline at Week 48 | 0.722 (17.7087) | 4.365 (16.0206)
  All participants, Change From Baseline at Week 96: number analyzed (Participants) | 56 | 53
  All participants, Change From Baseline at Week 96 | 3.274 (16.5408) | 1.625 (20.6684)

18. Secondary Outcome: Rate of Study Drug Compliance
Description: The rate of compliance was defined as the number of actual doses taken divided by the number of planned doses * 100. Participant-reported data were obtained from the participant's compliance log, which was completed by the participant or the caregiver. The participant or caregiver reported how many doses were taken. Compliance by drug accountability was determined by counting used and unused study drug sachets. All calculations were based on the records of the first dose date to the last dose date.
Time Frame: Baseline (Week 1 [Total Study Week 48]) up to EOT (Week 96 [Total Study Week 144])
Population: as for outcome 17
Measure: Median (Full Range); unit: percent of doses taken
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
percent of doses taken
  By drug accountability | 86.057 [27.03 to 106.06] | 80.118 [0 to 100.74]
  By participant-reported data: number analyzed (Participants) | 91 | 93
  By participant-reported data | 81.50 [0 to 99.9] | 78.59 [0 to 99.7]

19. Secondary Outcome: Predose Concentration of Ataluren
Description: Blood samples were drawn immediately before administration of the first daily dose (dose taken with breakfast) of ataluren. Whenever possible, the predose sample was to be obtained within 15 minutes of study ataluren administration.
Time Frame: Predose at Weeks 1, 16, 32, 48, 64, 80 and EOT (Week 96) (Total Study Weeks 48, 64, 80 96, 112, 128, and 144, respectively)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
micrograms/milliliter
  Week 1: number analyzed (Participants) | 6 | 7
  Week 1 | 1.668 (3.6279) | 0 (0)
  Week 16: number analyzed (Participants) | 90 | 90
  Week 16 | 5.744 (5.7198) | 7.552 (8.3963)
  Week 32: number analyzed (Participants) | 80 | 78
  Week 32 | 6.298 (7.1222) | 7.694 (7.9796)
  Week 48: number analyzed (Participants) | 78 | 69
  Week 48 | 5.874 (6.8533) | 6.981 (6.8874)
  Week 64: number analyzed (Participants) | 65 | 61
  Week 64 | 5.227 (4.7054) | 5.703 (6.2718)
  Week 80: number analyzed (Participants) | 58 | 59
  Week 80 | 6.126 (6.4939) | 4.902 (5.9218)
  Week 96: number analyzed (Participants) | 57 | 53
  Week 96 | 6.390 (6.8861) | 5.435 (6.5315)

20. Secondary Outcome: Number of Participants Who Required Interventions for Pulmonary Symptoms
Description: During treatment, any interventions including hospitalization or use of oral, inhaled, or IV antibiotics was documented if it was due to an exacerbation-like episode. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the Adverse Events module.
Time Frame: Baseline (Week 1 [Total Study Week 48]) up to EOT (Week 96 [Total Study Week 144])
Population: The Study 009e As-Treated Population: participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
Participants
  Hospitalization | 44 | 49
  Use of Inhaled Antibiotics | 10 | 18
  Use of Intravenous Antibiotics | 80 | 80

21. Secondary Outcome: Number of Participants With Disruptions in Activities of Daily Living Because of Pulmonary Symptoms
Description: During treatment, participants reported when they missed school or work because of pulmonary symptoms. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the Adverse Events module.
Time Frame: Baseline (Week 1 [Total Study Week 48]) up to EOT (Week 96 [Total Study Week 144])
Population: The Study 009e As-Treated Population: participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
Participants
  Missed at Least 1 Day of School | 23 | 25
  Missed at Least 1 Day of Work | 27 | 25

22. Secondary Outcome: Duration of Disruptions in Activities of Daily Living Because of Pulmonary Symptoms
Description: During treatment, participants reported when they missed school or work because of pulmonary symptoms. If Event Date was before Day 1 (Baseline) Date, Study Day = Event Date - First Dose Date. If Event Date was on or after Day 1 Date, Study Day = Event Date - First Dose Date + 1. The Duration = Return to Stable Date - Onset Date. Participants with a respiratory event that was ongoing when the participant was discontinued from the study were considered as not evaluable. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the Adverse Events module.
Time Frame: Baseline (Week 1 [Total Study Week 48]) up to EOT (Week 96 [Total Study Week 144])
Population: The Study 009e As-Treated Population: participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: days
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
days
  Missed at Least 1 Day of School | 25.0 [7 to 187] | 21.5 [4 to 112]
  Missed at Least 1 Day of Work | 25.0 [1 to 161] | 22.0 [1 to 131]

23. Secondary Outcome: Change From Baseline in Body Weight at Weeks 48 and 96
Description: Participants were weighed, and the weight was recorded at Baseline and then every 8 weeks during the treatment period. Baseline was Week 1. A positive change from Baseline indicates that weight increased.
Time Frame: Baseline (Week 1 [Total Study Week 48]), Week 48 (Total Study Week 96), EOT (Week 96 [Total Study Week 144])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
kilograms (kg)
  Baseline | 53.354 (13.5601) | 57.444 (11.7890)
  Change From Baseline at Week 48: number analyzed (Participants) | 78 | 70
  Change From Baseline at Week 48 | 1.232 (2.8322) | 0.540 (2.8287)
  Change From Baseline at Week 96: number analyzed (Participants) | 57 | 53
  Change From Baseline at Week 96 | 2.149 (5.0803) | 0.830 (3.6440)

24. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Weeks 48 and 96
Description: Participants were weighed and measured and the weight and height were recorded at each visit. The BMI was determined by dividing the participant's weight by his or her height. Baseline was Week 1. A positive change from Baseline indicates that BMI increased.
Time Frame: Baseline (Week 1 [Total Study Week 48]), Week 48 (Total Study Week 96), EOT (Week 96 [Total Study Week 144])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg/square meter (kg/m^2)
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 95 | 96
kg/square meter (kg/m^2)
  Baseline | 20.023 (3.3136) | 21.044 (2.7735)
  Change From Baseline at Week 48: number analyzed (Participants) | 78 | 70
  Change From Baseline at Week 48 | 0.179 (0.8323) | 0.102 (0.9179)
  Change From Baseline at Week 96: number analyzed (Participants) | 57 | 53
  Change From Baseline at Week 96 | 0.144 (1.1404) | 0.105 (1.1885)

25. Secondary Outcome: Total Lung Computed Tomography (CT) Score at Weeks 48 and 96
Description: Lungs were imaged by using non-contrast, spiral CT. The administration of CT scans was discontinued for this study via a memorandum sent to all Investigators, based on the results of Study 009, which showed that this exploratory endpoint failed to discriminate active treatment from placebo over the 48-week study period. Therefore, this Outcome Measure was removed from the study as a Secondary Outcome Measure and the CT scans that were administered for this study were not reviewed or analyzed for this Outcome Measure.
Time Frame: Week 48 (Total Study Week 96) and EOT (Week 96 [Total Study Week 144])
Population: The Study 009e As-Treated Population: participants who received at least 1 dose of study drug. Here, 'Number analyzed' signifies the number of participants analyzed for the specified weeks for this Outcome Measure.
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Change From Baseline in the Nasal Transepithelial Potential Difference (TEPD) at Week 48
Description: TEPD was to be assessed in each nostril by using standardized equipment, techniques, and solutions. Collection of nasal TEPD tracings was discontinued for this study via a memorandum sent to all Investigators, based on the results of Study 009, which showed that this biomarker failed to discriminate active treatment from placebo over the 48-week study period. Therefore, this Outcome Measure was removed from the study as a Secondary Outcome Measure and none of the nasal TEPD tracings were reviewed or analyzed for this Outcome Measure.
Time Frame: Baseline (Week 1 [Total Study Week 48]) and Week 48 (Total Study Week 96)
Population: as for outcome 25
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Change From Baseline in the Concentration of Sweat Chloride at Week 48
Description: Sweat was collected, from each arm, by using pilocarpine iontophoresis. The chloride concentration in the sweat was quantified for each arm by using standard laboratory methods. Tests were considered valid if the sweat collection time was ≤35 minutes; tests with longer collection times were also considered valid if extra time was needed to obtain sufficient volume (≥15uL) for analysis. For analysis purposes, the average of the values from each arm were computed. If the assessment was valid and/or available in only 1 arm, this value was used as if it were the average of both arms. The method used was consistent with the guidelines of the Cystic Fibrosis Foundation Therapeutics - Therapeutic Development Network. Baseline was the most recent value of sweat chloride prior to treatment in Study 009e. A positive change from Baseline indicates that sweat chloride concentration increased.
Time Frame: Baseline (Week 1 [Total Study Week 48]), Week 48 (Total Study Week 96)
Population: The Study 009e As-Treated Population: participants who received at least 1 dose of study drug. Here, 'Number Analyzed' signifies participants evaluable for the specified week. One and 4 participants in the ataluren/ataluren and placebo/ataluren groups, respectively, were not evaluable.
Measure: Mean (Standard Deviation); unit: millimoles/liter
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren
Number analyzed (Participants) | 94 | 92
millimoles/liter
  Baseline | 100.26 (13.602) | 97.88 (16.444)
  Change From Baseline at Week 48: number analyzed (Participants) | 48 | 41
  Change From Baseline at Week 48 | 5.34 (10.062) | 3.60 (14.422)

ADVERSE EVENTS:
Time Frame: Baseline (Week 1 [Total Study Week 48]) up to 4 Weeks Post-Treatment (Week 100 [Total Study Week 148]) or PD (whichever occurred first)
Description: The Study 009e As-Treated Population: participants who received at least 1 dose of study drug.
Groups:
- Overall Population: Participants who received double-blind ataluren or placebo during Study 009 received open-label ataluren TID: 10 mg/kg of body weight with breakfast, 10 mg/kg with lunch, and 20 mg/kg with dinner (total dose 40 mg/kg/day), for up to 96 weeks. Participants were followed for 4 weeks after treatment.
Arm/Group | Ataluren/Ataluren | Placebo/Ataluren | Overall Population
Serious Adverse Events (participants affected / at risk) | 48/95 | 57/96 | 105/191
Other Adverse Events (participants affected / at risk) | 95/95 | 94/96 | 189/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ataluren/Ataluren (N=95) | Placebo/Ataluren (N=96) | Overall Population (N=191)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Annual fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (3)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (2) | 1 (1) | 2 (3)
Mycobacterium abscessus infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Burkholderia cepacia infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Catheter sepsis (Infections and infestations) | 1 (2) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Hypercreatininaemia (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Nephritis interstitial (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Cystic fibrosis lung (Respiratory, thoracic and mediastinal disorders) | 41 (84) | 45 (90) | 86 (174)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 1 (1) | 3 (7)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (2)
Axillary vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren/Ataluren (N=95) | Placebo/Ataluren (N=96) | Overall Population (N=191)
Diarrhoea (Gastrointestinal disorders) | 13 | 16 | 29
Abdominal pain (Gastrointestinal disorders) | 14 | 13 | 27
Constipation (Gastrointestinal disorders) | 12 | 15 | 27
Vomiting (Gastrointestinal disorders) | 9 | 13 | 22
Abdominal pain upper (Gastrointestinal disorders) | 8 | 13 | 21
Nausea (Gastrointestinal disorders) | 5 | 16 | 21
Abdominal distension (Gastrointestinal disorders) | 5 | 4 | 9
Pyrexia (General disorders) | 19 | 19 | 38
Fatigue (General disorders) | 4 | 13 | 17
Drug hypersensitivity (Immune system disorders) | 2 | 7 | 9
Viral upper respiratory tract infection (Infections and infestations) | 26 | 32 | 58
Rhinitis (Infections and infestations) | 13 | 15 | 28
Nasopharyngitis (Infections and infestations) | 13 | 14 | 27
Sinusitis (Infections and infestations) | 11 | 13 | 24
Respiratory tract infection bacterial (Infections and infestations) | 9 | 10 | 19
Lung infection pseudomonal (Infections and infestations) | 11 | 7 | 18
Pharyngitis (Infections and infestations) | 6 | 10 | 16
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 6 | 6 | 12
Bronchitis (Infections and infestations) | 6 | 5 | 11
Bronchopulmonary aspergillosis (Infections and infestations) | 6 | 5 | 11
Respiratory tract infection fungal (Infections and infestations) | 6 | 3 | 9
Upper respiratory tract infection (Infections and infestations) | 3 | 6 | 9
Oral fungal infection (Infections and infestations) | 2 | 5 | 7
Pulmonary function test decreased (Investigations) | 9 | 3 | 12
Abnormal loss of weight (Metabolism and nutrition disorders) | 2 | 9 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 10 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 8 | 14
Headache (Nervous system disorders) | 12 | 14 | 26
Insomnia (Psychiatric disorders) | 1 | 6 | 7
Anxiety (Psychiatric disorders) | 1 | 5 | 6
Hypercreatininaemia (Renal and urinary disorders) | 7 | 9 | 16
Dysuria (Renal and urinary disorders) | 4 | 9 | 13
Cystic fibrosis lung (Respiratory, thoracic and mediastinal disorders) | 66 | 69 | 135
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 28 | 57
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 13 | 18 | 31
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 11 | 19
Rales (Respiratory, thoracic and mediastinal disorders) | 10 | 9 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 16
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 10
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 6
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 5
Rash (Skin and subcutaneous tissue disorders) | 3 | 8 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 7 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.